CLINICAL TRIAL: NCT03470038
Title: The Interaction Between NGF-induced Muscle Sensitivity and Acute Exercise-induced Ischemia
Brief Title: Interaction Between NGF and Acute Exercise-induced Ischemia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Line Bay Sørensen, PhD. stud., Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: N-2017-0007_S2
Record Dates: First submitted 2018-03-13; First posted 2018-03-19 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Hyperalgesia; Pain Response; Healthy Subjects
Keywords: NGF-induced pain; Ischemia-induced pain; Hyperalgesia; NGF pain model
MeSH Terms: conditions — Hyperalgesia | interventions — Nerve Growth Factor; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NGF condition + Control condition (Experimental): All participants will receive five injections with NGF (1ug/0.5ml) into the tibialis anterior muscle in their non-dominant leg
  After 4 weeks:
  All participants will receive five injections with isotonic saline (9%/0.5ml) into the tibialis anterior muscle in their non-dominant leg
  Interventions: Drug: NGF; Drug: Isotonic saline
- Control condition + NGF condition (Experimental): All participants will receive five injections with isotonic saline (9%/0.5ml) into the tibialis anterior muscle in their non-dominant leg
  After 4 weeks:
  All participants will receive five injections with NGF (1ug/0.5ml) into the tibialis anterior muscle in their non-dominant leg
  Interventions: Drug: NGF; Drug: Isotonic saline

INTERVENTIONS:
Drug: NGF — Intramuscular injection
  Other Names: Beta-Nerve Growth Factor, Human
Drug: Isotonic saline — Intramuscular injection
  Other Names: Control

SUMMARY:
The purpose of this study is to investigate pain evoked responses and facilitation of NGF-induced mechanical muscle hyperalgesia over time following an acute exercised-induced ischemic condition in a NGF-sensitized muscle.

DETAILED DESCRIPTION:
Assessing evoked pain responses and muscle hyperalgesia following contractions during acute ischemia in a NGF-sensitized muscle may clarify whether an interaction between NGF sensitization and acidic stimulation exist.

It is hypothesized that acute ischemic exercise with the NGF-sensitized TA muscle, in contrast to ischemic exercise in a non-sensitized would: 1) potentiate pain-evoked responses, and 2) facilitate NGF-induced muscle hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and pain free volunteers

Exclusion Criteria:

* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, mental illnesses, or psychiatric diseases.
* Past history of chronic pain in the musculoskeletal system (muscle, joint, cartilage, connective tissue)
* Participation in other pain trials throughout the study period
* Lack of ability to cooperate
* Taking any analgesic 24 hours before the injections
* Performing any strenuous leg exercise through out the study period causing sore muscles

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Muscle sensitivity | Change from baseline at 1 week
  Pressure pain thresholds (PPTs) are assessed over the non-dominant tibialis anterior muscle using a handhold pressure algometer.

SECONDARY OUTCOMES:
Ischemic-induced pain intensity | Assessed right after the dorsiflexions have been performed
  Subjects perform 45 dorsiflexions with their non-dominant leg while a cuff is mounted over the knee to occlude the blodflow from the muscle (ischemia) Subjects subsequently rate their perceived pain intensity verbally on a numeric rating scale (NRS)
Functional muscle pain | Change from baseline at 1 week
  Subjects evaluate their muscle pain during movement using a Likert Scale for lower limp
Muscle pain diary | Change from baseline at 1 week
  Subjects evaluate their muscle pain during movement using a Likert Scale for lower limp and perceived pain intensity at rest on a numeric rating scale (NRS). The diary is filled out at home on days between sessions

CONTACTS AND LOCATIONS:
Overall Officials: Line Bay Sørensen, Ph.d stud., Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorensen LB, Gazerani P, Graven-Nielsen T. Nerve growth factor-induced muscle hyperalgesia facilitates ischaemic contraction-evoked pain. Eur J Pain. 2019 Nov;23(10):1814-1825. doi: 10.1002/ejp.1455. Epub 2019 Aug 5. PMID 31314952